CLINICAL TRIAL: NCT02388750
Title: Prospective Study of Palonosetron in the Prophylaxis/Rescue of Radiation Induced Nausea and Vomiting (RINV) - a Phase II Study
Brief Title: Prospective Study of Palonosetron in Radiation Induced Nausea and Vomiting (RINV)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dr. Edward Chow (Other)
Responsible Party: Sponsor-Investigator, Dr. Edward Chow, Professor, Sunnybrook Health Sciences Centre
Organization: Sunnybrook Health Sciences Centre (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Palonosetron
Record Dates: First submitted 2015-02-20; First posted 2015-03-17 (Estimated); Last update posted 2017-10-06 (Actual); Status verified 2017-10

CONDITIONS: Nausea; Vomiting
Keywords: nausea; vomiting; radiation; anti-emetic drug
MeSH Terms: conditions — Nausea; Vomiting | interventions — Palonosetron

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- No previous nausea and vomiting (Other): Palonosetron 0.5 mg oral capsule given for the length of radiation treatment
  No previous nausea and vomiting 24 hours prior to radiotherapy
  Interventions: Drug: Palonosetron; Radiation: Low or moderate risk radiotherapy
- Previous nausea and/or vomiting (Other): Palonosetron 0.5 mg oral capsule given for the length of radiation treatment
  Previous nausea and/or vomiting 24 hours prior to radiotherapy
  Interventions: Drug: Palonosetron; Radiation: Low or moderate risk radiotherapy

INTERVENTIONS:
Drug: Palonosetron — Palonosetron 0.5 mg every other day until completion of radiation and at least one hour prior on days of RT
Radiation: Low or moderate risk radiotherapy — Low or moderately emetogenic radiotherapy will be given to all patients on study.

SUMMARY:
This phase II study will investigate the use of palonosetron in the efficacy of prophylaxis or rescue of single or multiple fraction radiation induced nausea and vomiting. This prospective study employs a parallel arm design, allowing for inclusion of patients with pre-existing nausea and vomiting versus no current nausea or vomiting. Eligible patients receiving radiotherapy known to have a low or moderate emetogenic risk will receive every other day dosing of 0.5 mg palonosetron for the length of treatment. Nausea, vomiting, use of rescue medication, and impact on quality of life will be monitored during and after radiation treatment completion.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent
* Patient will receive radiation therapy to considered moderate risk (upper abdomen, upper and half body irradiation) or low risk (lower thorax and pelvis) emetogenic palliative radiotherapy.
* Patients will be grouped according to nausea and vomiting status at baseline as follows:

  * Group 1: Patient is experiencing no nausea and vomiting at baseline
  * Group 2: Patient is experiencing at least mild nausea and/or at least mild vomiting at baseline

Exclusion Criteria:

* Patient is scheduled to receive cranial radiation therapy during or within 10 days following completion of protocol RT.
* Patient received cranial RT within 7 days prior to commencement of protocol RT.
* Patient is scheduled to receive chemotherapy during or within 10 days following completion of protocol RT.
* Patient received moderately or highly emetogenic chemotherapy within 7 days prior to commencement of protocol RT.
* Patient is scheduled to change regimen/dose or start the use of low dose corticosteroids (inhaled or topical permitted), or other medications considered to have antiemetic properties within 48 hours prior to protocol RT.
* Patient is scheduled to change regimen/dose or start the use of low dose corticosteroids (inhaled or topical permitted), or other medications considered to have antiemetic properties during or within 10 days following completion of protocol RT.
* Concurrent use of corticosteroids during protocol RT is not permitted, unless low dose corticosteroids (hydrocortisone) are used for cancer treatment
* Patient is allergic to protocol medication.
* Patient has a Karnofsky Performance Status score <40.
* Patient is a woman who is pregnant or of childbearing potential and is not using contraceptive measures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2015-04; Primary Completion 2017-08-07 (Actual); Study Completion 2017-08-07 (Actual)

PRIMARY OUTCOMES:
Efficacy for prevention of nausea and vomiting events as measured by a daily diary | Day 0 to Day 10 post-radiation
  Primary outcome is to determine the efficacy of palonosetron for the prevention of radiation-induced vomiting in patients undergoing low or moderate emetogenic radiation therapy. Daily diary collects events of nausea and/or vomiting, and corresponding severity.

SECONDARY OUTCOMES:
Complete prophylaxis of nausea | Day 0 to Day 10 post-radiation
  Proportion of patients achieving complete prophylaxis of nausea and not requiring the use of any, or supplemental rescue antiemetic medication during and in the 10 days following radiation therapy
Complete prophylaxis of vomiting | Day 0 to Day 10 post-radiation
  Proportion of patients achieving complete prophylaxis of vomiting without requiring the use of any, or supplemental rescue antiemetic medication during and in the 10 days following radiation therapy
Partial control of nausea | Day 0 to Day 10 post-radiation
  Proportion of patients achieving partial control of nausea during and in the 10 days following radiation therapy
Partial control of vomiting | Day 0 to Day 10 post-radiation
  Proportion of patients achieving partial control of vomiting during and in the 10 days following radiation therapy
Time to use of rescue medication | Day 0 to Day 10 post-radiation
  Median time from first fraction of radiation therapy to first use or increase in use of rescue medication
Time to nausea | Day 0 to Day 10 post-radiation
  Median time from first fraction of radiation therapy to first episode or increase in episodes of nausea
Time to vomiting | Day 0 to Day 10 post-radiation
  Median time from first fraction of radiation therapy to first episode or increase in episodes of vomiting
Quality of life | Baseline, during the 5th and 10th day of radiation (if applicable), and 3, 5, 7, and 10 days post radiation.
  Quality of life as measured by the EORTC QLQ-C15-PAL and the FLIE.
Adverse effects | Day 0 to Day 10 post-radiation
  The side effects of constipation and headache will be monitored throughout the study period graded according to the CTCAE criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Chow Edward, MBBS PhD, Principal Investigator — Odette Cancer Centre, Sunnybrook Health Sciences Centre
Locations (1):
- Odette Cancer Centre, Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada